CLINICAL TRIAL: NCT02524080
Title: Healthcare at Optimal Care Level for Patients Who Needs Primary Care - Collaboration Between Care Providers From The Emergency Medical Services' Perspective
Brief Title: Healthcare at Optimal Care Level for Patients Who Needs Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Boras (Other)
Responsible Party: Principal Investigator, Birgitta Wireklint Sundström, Birgitta Wireklint Sundström, RNAN, PhD (Associate professor), University of Boras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBoras
Record Dates: First submitted 2015-08-11; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Patients Compliance
Keywords: Ambulance; Trust; Patients; Healthcare chain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Emergency Department (Other): Triage to optimal healthcare level
  Interventions: Procedure: Triage to optimal healthcare level
- Healthcare Center (Other): Triage to optimal healthcare level
  Interventions: Procedure: Triage to optimal healthcare level

INTERVENTIONS:
Procedure: Triage to optimal healthcare level — Triage to optimal healthcare level

SUMMARY:
If patients get to optimal level of healthcare directly it will prevent suffering for both patients and their relatives and moreover save a lot of resources. In the project "Care at the right care level" (CRC) the Emergency Medical Services (EMS) will triage patients who are in need of primary health care to the Primary Care (PC) instead of to the Emergency Department (ED). This intervention should be implemented with the same medical safety as with traditional care in the ED and the patient and their relatives should experience corresponding confidence to the healthcare provider. To prepare this intervention this patient group and their care needs have to be identified by a retrospective journal review and a guideline has to be developed. To evaluate the patients' and their relatives' experience of the intervention, finally interviews will be implemented. This project is expected to provide answers whether it is possible to triage non-urgent patients to another care level with the same medical safety and that the patients experience the same confidence in healthcare. And further it will answer the question, if the care providers around the patient manage to collaborate.

DETAILED DESCRIPTION:
Background

The research has a caring science approach, which has the patient in focus, with the general aim to describe care that strengthens and supports health. Further, a health care science approach recognizes the patient's suffering as a motivation for care.

In this study a non-urgent patient is a patient with illness, injury or ill-health suitable for the health care received in PC. The PC is able to take care of problems that not urgent and unlikely to require admission. The problem should not need specialized service in an ED, such as facilities, urgent intervention, rapid and/or complex diagnostic and could equally be managed at the PC.

For increased survival, reduced risk of complications and ability to quickly return to a functional life, it is important that there is a coherent chain of care. The EMS with the Prehospital Emergency Nurses (PEN:s) is an important part of many treatment chains, fast tracks and pathways, for example for patients with stroke, heart attack, hip fracture and geriatric care.The care model the EMS currently follows, means that virtually all patients transported to ED regardless of medical need and seriousness, which is consistent with current medical guidelines. Studies shows that around 25 % of patients arriving to the ED should have been treated at another level of care for having the right care. There is also a connection between increased mortality and overloading in the ED.

The need for emergency care is large and tends to increase, particularly in the elderly population (≥ 65 years). For resources to be utilized effectively, the health care has to be given at the level of care that is most appropriate. This requires that different providers that all have a responsibility for the patients can think outside the box, based on the individual patient's need of care. In addition, assumes cooperation and coordination to enable organizational change, which can provide good care from the patient's perspective.

The numbers of care seekers tend to rise and health care resources must be used more efficiently to cope with the increasing patients. Today the healthcare providers, the Country Council, the PC and Community Care, don't collaborate with each other, although they all have a shared responsibility. According to health care prioritization decisions, witch control the need of care and time to care. For resources to be utilized efficiently, care is provided at the care level that is most appropriate. However this cannot be achieved today, because of the regional guidelines.

The problem exists nationally and studies show that it is also an internationally problem, and as the number of care seekers increases, the problem tends to grow. Studies explain that a lot of patients could go to the PC. And some means that one third of the patients should have their care at another level than ED.

A new model with extended prehospital emergency care, which not has been tried before, means that assessment of the patient's condition and the need for continuing care is made at collection point, if the patient's medical condition make this possible. The health care model called "Care at the right care level" (CRC), means that the assessment and treatment interventions are implemented, and decisions on further treatment is planned in consultation with the general physician (GP) in the patient's PC. Decisions on continuing care can, for example, implicate that the patient receives a visit time to the GP immediately or later, or run directly to the ED.

Aims The overall aim is to investigate if it is possible for the Prehospital Emergency Nurse (PEN) to triage non-urgent patients to optimal care level in the the Primary Care (PC).

Issues:

* How do patients experience trust to the healthcare?
* Is the new care model medical safe?

Study 1

Title: Swedish emergency medical services' identification of potential candidates for primary healthcare. Resubmitted June 2015, Scandinavian Journal of Primary Health Care.

The aim is to investigate if it is possible to isolate and identify the patient group and their care needs, which can be triaged at the primary care instead of to the ED.

Study 2

Title: Patients with suspected primary healthcare problems using the emergency medical services - Developing a questionnaire to measure patient trust in healthcare. In manuscript.

The aim is to developing an instrument for measuring patient's confidence to the health care.

Study 3

Title: Care at the right care level - an intervention study. Ongoing from April 2013.

The aim of the study is to investigate if it is possible to triage less sick or injured patients to another level of care with the same medical safety and that they still have the same confidence to the healthcare.

Study 4

Title: Prehospital emergency care for patients with primary care needs - Patients' experiences

The aim of the study is to describe the patient's lived experiences of being treated in the new caring model.

Ethical considerations

In the interventions study (study 3), there will be a risk that the patient need a secondary transport from the Healthcare Center to the ED. To reduce that risk the PEN always take a contact with the physician at the Primary care clinic, when the patient in the CRC-project is randomized to The Primary care. It is also always a risk that the patient feels depended and feels duty to participate in the study. So it is important that the PEN provides correct information about the free will. Except the above mentioned ethical considerations no other are aspected to arise. The benefit is considered high, while the risk is considered small.

Hypothesis

With the CRC-model the patients receive optimal health care and feel the same trust to the healthcare as the traditional healthcare.

Primary and secondary endpoints.

The primary endpoint is the proportion who received optimal care and experiencing the same trust in the care than to the traditional care.Secondary endpoints are correct preliminary assessment/final diagnosis without secondary transport.

The relation between the studies is logical. To do an intervention study, it is necessary to know witch patient´s is possible to include. And the PEN needs a decision support for their help to triage right patient to right level of care (study 1). For evaluating if patients still feel the same confidence to the healthcare, a measuring instrument is needed, and it also has to be validated (study 2). To know if it is possible to triage the non-urgent patient group to the Healthcare Center, the investigators have to try the intervention, and evaluate the project (study 3). To get a deeper understanding for the patients and his relatives experiences of obtaining the new healthcare model, interviews will be done (study 4).

ELIGIBILITY:
Inclusion Criteria:

* Un-urgent patient in ambulance
* Age from 18 years
* No communication problems
* No dementia or disorientation
* Not in need of special examinations

Exclusion Criteria:

* No

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-06 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
To measure patient trust in healthcare - Questionnaire | 2-3 days
  A lickert scale with possible responses as follows (scores in parentheses): strongly disagree (1), disagree (2), neither disagree nor agree (3), agree (4) and strongly agree (5).

CONTACTS AND LOCATIONS:
Overall Officials: Johan Herlitz, Professor, Study Director — University of Boras, Sweden